CLINICAL TRIAL: NCT00264524
Title: DNA Typing of HLA-DR/DQ Alleles in Taiwan Chinese With Rheumatic Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Allocation: Non-Randomized | Masking: None | Purpose: Diagnostic
Other Study IDs: CMU93-M-34
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2004-01

CONDITIONS: Rheumatic Heart Disease
Keywords: Rheumatic heart disease, HLA, Genetics, Taiwan
MeSH Terms: conditions — Rheumatic Heart Disease

INTERVENTIONS:
Procedure: venipuncture to withdraw patient's blood

SUMMARY:
The current study was designed to determine whether the HLA-DRB1, DQA1, DQB1 alleles are associated with the risk and the pattern of valve damage of RHD.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients with Rheumatic mitral stenosis 2.Chinese Han ethnicity

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult
Dates: Start 2004-01; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Tai Chou, MD, PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- Division of cardiology, China Medical University Hospital, Taichung, Taiwan